CLINICAL TRIAL: NCT04653909
Title: The Effectiveness of Rehabilitation Program in an Ultra-rare Calfan Syndrome
Brief Title: The Physiotherapy and Rehabilitation in Calfan Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant of professeur, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/032
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: CALFAN Syndrome
Keywords: ataxia; rehabilitation; disabilities
MeSH Terms: conditions — Ataxia | interventions — Rehabilitation; Orthotic Devices

STUDY DESIGN:
Intervention Model Description: Case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case (Experimental): A patient who was diagnosed with the calfan syndrome
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The abdominal and back strengthening exercises on the mat, the open-closed perturbation training in sitting and standing positions for trunk control. Functional exercises were performed in the same positions for simulating daily living activities. The stretching and strengthening exercises were applied to her scoliosis and also given trunk orthoses.
  Other Names: Orthoses

SUMMARY:
Calfan syndrome is a progressive neurodegenerative systemic disease. It is a rare and difficult disease to diagnose due to the complex symptoms that occur over the years to postpartum. The aim of this study is to investigate the effectiveness of the physiotherapy and rehabilitation program in a rare case with Calfan syndrome.

DETAILED DESCRIPTION:
13 years old, a female patient was diagnosed with Calfan syndrome one year ago. Only 11 patients have been identified in the literature. Its phenotype is characterized by recurrent episodes of liver failure and hepatic fibrosis in early childhood. Our patient had neurological symptoms that were gait disturbances, ataxia and tremor, as well as peripheral neuropathy and cognitive impairment. Also, musculoskeletal problems such as scoliosis, hip dysplasia, osteoporosis, thoracic kyphosis, and increased lordosis were observed.

ELIGIBILITY:
Inclusion Criteria:

* Calfan syndrome

Exclusion Criteria:

* Any surgery in past six months

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Trunk Control | 3 month
  The Trunk Disorder Scale (TIS) was used to assess static and dynamic sitting balance and trunk coordination
The severity of ataxia | 3 month
  The International Ataxia Rating Scale (ICARS) was used to determine the severity
The quality of life | 3 month
  The Children's Quality of Life Scale (PedsQL) was used determine to quality of life level.
The Functional Independence | 3 month
  The Functional Independence Scale for Children (WeeFIM) was used determine to independence level.

SECONDARY OUTCOMES:
Upper extremity functional performance | 3 month
  The 9-Hole Peg test was used to evaluate upper extremity performance
Upper extremity disability level | 3 month
  the Quick Questionnaire for Arm, Shoulder and Hand Problems (Q-DASH) scale was used to evaluate physical disability and symptoms of upper extremity

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The applied rehabilitation protocol.
Supporting Information: CSR
Time Frame: Five years

REFERENCES:
- [Background] Spagnoli C, Frattini D, Salerno GG, Fusco C. On CALFAN syndrome: report of a patient with a novel variant in SCYL1 gene and recurrent respiratory failure. Genet Med. 2019 Jul;21(7):1663-1664. doi: 10.1038/s41436-018-0389-6. Epub 2018 Dec 10. No abstract available. PMID 30531813
- [Background] Lenz D, McClean P, Kansu A, Bonnen PE, Ranucci G, Thiel C, Straub BK, Harting I, Alhaddad B, Dimitrov B, Kotzaeridou U, Wenning D, Iorio R, Himes RW, Kuloglu Z, Blakely EL, Taylor RW, Meitinger T, Kolker S, Prokisch H, Hoffmann GF, Haack TB, Staufner C. SCYL1 variants cause a syndrome with low gamma-glutamyl-transferase cholestasis, acute liver failure, and neurodegeneration (CALFAN). Genet Med. 2018 Oct;20(10):1255-1265. doi: 10.1038/gim.2017.260. Epub 2018 Feb 8. PMID 29419818
- [Background] Lenz D, Staufner C, Wachter S, Hagedorn M, Ebersold J, Gohring G, Kolker S, Hoffmann GF, Jung-Klawitter S. Generation of an induced pluripotent stem cell (iPSC) line, DHMCi005-A, from a patient with CALFAN syndrome due to mutations in SCYL1. Stem Cell Res. 2019 May;37:101428. doi: 10.1016/j.scr.2019.101428. Epub 2019 Mar 22. PMID 30959346